CLINICAL TRIAL: NCT03367221
Title: Physiological Response to Different Levels of Support in Lung Transplant Recipients Undergoing Neurally Adjusted Ventilatory Assist (NAVA)
Brief Title: Physiological Response in Lung Transplant Recipients Undergoing Neurally Adjusted Ventilatory Assist
Acronym: TRANS-NAVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Prof, Policlinico Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRANS-NAVA
Record Dates: First submitted 2017-11-24; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Work of Breathing; Lung Transplant; Complications; Neurally Adjusted Ventilatory Assist; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAVA group (Experimental): NAVA ventilation
  Interventions: Device: NAVA ventilation

INTERVENTIONS:
Device: NAVA ventilation — Assisted Ventilation Mode, synchronized, through EAdi catheter, with patient's inspiratory effort and proportional to respiratory drive

SUMMARY:
Primary Graft Dysfunction (PGD) respresents the leading cause of mortality in early post-operative period of Lung Tranplantation (LTx). Protective ventilatory strategy could potentially reduce the risk of PGD in these patients. Neurally Adjusted Ventilatory Assist (NAVA) is an assisted ventilation mode that could allow to adopt this strategy. Aim of the study is to assess the feasibility of NAVA in the early post-LTx phase and to describe the breathing pattern and the physiological relationship between neural respiratory drive and different levels of ventilatory assist, in the absence of pulmonary vagal afferent feedback.

DETAILED DESCRIPTION:
Lung transplantation (LTx) is an important treatment option for select patients with end-stage pulmonary disease. Primary Graft Dysfunction (PGD) is the main cause of death; in the early period following LTx a protective ventilatory strategy (tidal volume - Vt of 6 mL/Kg + Positive End Expiratory Pressure) could potentially reduce the risk of PGD in these patients. Neurally Adjusted Ventilatory Assist (NAVA) is an assisted ventilation mode in which neural inspiratory activity is monitored through the continuous recording of electrical activity of the diaphragm (EAdi). Actually, Guidelines about the adoption of a protective ventilatory strategy in the early post-opeartive period are lacking.

NAVA, because of its intrinsic properties (proportionality between respiratory drive and level of assist, prevention of diaphragm atrophy), could allow to reach the afore mentioned ventilatory strategy. So, aim of the study, is the evaluation of patients' neural breathing pattern during NAVA, in early post-operative period of LTx

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y.o.
* Admission to ICU for post-operative monitoring after LTx
* Presence of spontaneous breathing activity
* Sedation titrated to a target RASS between 0 and -2
* Written informed consent obtained

Exclusion Criteria:

* Contraindication to nasogastric tube insertion (gastroesophageal surgery in the previous 3 months, gastroesophageal bleeding in the previous 30 days, history of esophageal varices, facial trauma)
* Increased risk of bleeding with nasogastric tube insertion, due to severe coagulation disorders and severe thrombocytopenia ( i.e., INR > 2 and platelets count < 70.000/mm3)
* Severe hemodynamic instability (noradenaline > 0.3 μg/kg/min and/or use of vasopressin)
* Postoperative extracorporeal respiratory support (ECMO)
* Pre-operative reconditioning of the transplanted lungs by means of ex-vivo lung perfusion (EVLP)
* Lung retransplantation
* Failure to obtain a stable EAdi signal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the variations of Electrical Activity of the Diaphragm in response to different levels of ventilatory assist at different degrees of lung inflation (different Positive End Expiratory Pressure values) | One hour after the recovery of spontaneous breathing
  Electrical Activity of the Diaphragm (EAdi) (microVolt)
Evaluation of the variations of Neuro-Mechanical Coupling (expressed as microVolt of EAdi /cmH2O of airway pressure Ratio) in response to different levels of ventilatory assist at different degrees of lung inflation | One hour after the recovery of spontaneous breathing
  Neuro-Mechanical Coupling (NMC) (microvolt/cmH2O)
Evaluation of the variations of Neuro-ventilatory Efficiency (expressed as microvolt of EAdi / mL of Tidal Volume Ratio) in response to different levels of ventilatory assist at different degree of lung inflation | One hour after the recovery of spontaneous breathing
  Neuro-Ventilatory Efficiency (NVE) (microvolt/mL)
Evaluation of the changes in the patient's neural breathing pattern (expressed as mL of Tidal Volume) at different levels of ventilatory assist | One hour after the recovery of spontaneous breathing
  Tidal Volume (mL)
Evaluation of the changes in the patient's neural breathing pattern (expressed as respiratory rate) at different levels of ventilatory assist | One hour after the recovery of spontaneous breathing
  Respiratory rate (Breaths/min)

SECONDARY OUTCOMES:
Evaluation of the feasibility of Plateau Pressure during NAVA | One hour after the recovery of spontaneous breathing, with inspiratory hold manoeuvres
  Plateau Pressure (Pplat)
Ultrasound assessment of the changes of Diaphragm's Thickening Fraction at different levels of Positive End Expiratory Pressure and at different NAVA gains | One hour after the recovery of spontaneous breathing
  Diaphragm's Thickening Fraction (TF)
Assesment of the total asynchrony index (double triggering + missed efforts + inspiratory trigger delay +short cycling + prolonged cycling) | One hour after the recovery of spontaneous breathing
  Total Asinchrony Index

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Abbruzzese, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Luigi Castagna, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Nicola Bottino, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Alberto Zanella, MD, Principal Investigator — University of Milan; Nadia Corcione, MD, Principal Investigator — Fondazione IRCCS Ca' Granda; Antonio Pesenti, Prof, Principal Investigator — University of Milan
Locations (2):
- Ospedale Maggiore Policlinico, Milan, Italy
- University Hospital of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grasselli G, Castagna L, Abbruzzese C, Corcione N, Bottino N, Guzzardella A, Colombo SM, Carlesso E, Mauri T, Rossetti V, Palleschi A, Scaravilli V, Zanella A, Pesenti A. Pulmonary volume-feedback and ventilatory pattern after bilateral lung transplantation using neurally adjusted ventilatory assist ventilation. Br J Anaesth. 2021 Jul;127(1):143-152. doi: 10.1016/j.bja.2021.03.010. Epub 2021 Apr 21. PMID 33892948